CLINICAL TRIAL: NCT01459588
Title: Safety, Efficacy, and Acceptability Study of an Eye Drop Formulation in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10146X-001
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Carboxymethylcellulose Based Eye Drop Formulation A (Experimental): Carboxymethylcellulose Based Eye Drop Formulation A (Refresh Optive® Advanced Sensitive Eye Drops) 1-2 drops in each eye as needed, at least 2 times daily for 30 days.
  Interventions: Drug: Carboxymethylcellulose Based Eye Drop Formulation A
- Carboxymethylcellulose Based Eye Drop Formulation B (Experimental): Carboxymethylcellulose Based Eye Drop Formulation B (Refresh Optive® Advanced Eye Drops) 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Interventions: Drug: Carboxymethylcellulose Based Eye Drop Formulation B
- Carboxymethylcellulose Preservative-Free Lubricant Eye Drops (Active Comparator): Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops (Optive® Sensitive Preservative-Free Lubricant Eye Drops) 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Interventions: Drug: Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops
- Carboxymethylcellulose Based Lubricant Eye Drops (Active Comparator): Carboxymethylcellulose Based Lubricant Eye Drops (Optive® Lubricant Eye Drops) 1-2 drops in each eye as needed, at least 2 times daily for 30 days.
  Interventions: Drug: Carboxymethylcellulose Based Lubricant Eye Drops

INTERVENTIONS:
Drug: Carboxymethylcellulose Based Eye Drop Formulation A — Carboxymethylcellulose Based Eye Drop Formulation A (Refresh Optive® Advanced Sensitive Eye Drops) 1-2 drops in each eye as needed, at least 2 times daily for 30 days.
  Other Names: Refresh Optive® Advanced Sensitive Eye Drops
  Arms: Carboxymethylcellulose Based Eye Drop Formulation A
Drug: Carboxymethylcellulose Based Eye Drop Formulation B — Carboxymethylcellulose Based Eye Drop Formulation B (Refresh Optive® Advanced Eye Drops) 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Other Names: Refresh Optive® Advanced Eye Drops
  Arms: Carboxymethylcellulose Based Eye Drop Formulation B
Drug: Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops — Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops (Optive® Sensitive Preservative-Free Lubricant Eye Drops) 1-2 drops in each eye as needed at least 2 times daily for 30 days.
  Other Names: Optive® Sensitive Preservative-Free Lubricant Eye Drops
  Arms: Carboxymethylcellulose Preservative-Free Lubricant Eye Drops
Drug: Carboxymethylcellulose Based Lubricant Eye Drops — Carboxymethylcellulose Based Lubricant Eye Drops (Optive® Lubricant Eye Drops) 1-2 drops in each eye as needed, at least 2 times daily for 30 days.
  Other Names: Optive® Lubricant Eye Drops
  Arms: Carboxymethylcellulose Based Lubricant Eye Drops

SUMMARY:
This study will evaluate the safety, efficacy, and acceptability of an eye drop formulation in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Dry eyes
* Current use of eye drops for dry eye at least twice daily, on average for at least 3 months

Exclusion Criteria:

* Cataract, laser-assisted in situ keratomileusis (LASIK), or photorefractive keratectomy (PRK) surgery in the last 12 months
* Need to wear contact lenses during the study, or has worn contact lenses in the last 6 months
* Active ocular allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2012-02-15 (Actual); Study Completion 2012-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Petaluma, California, United States

REFERENCES:
- [Background] Simmons PA, Carlisle-Wilcox C, Vehige JG. Comparison of novel lipid-based eye drops with aqueous eye drops for dry eye: a multicenter, randomized controlled trial. Clin Ophthalmol. 2015 Apr 15;9:657-64. doi: 10.2147/OPTH.S74849. eCollection 2015. PMID 25931806

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Started | 105 | 51 | 103 | 56
Completed | 104 | 49 | 102 | 55
Not Completed | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops | Total
Number analyzed (Participants) | 105 | 51 | 103 | 56 | 315
Age, Customized [Number; unit: Participants]
  <30 years | 9 | 5 | 6 | 5 | 25
  30 to 40 years | 10 | 3 | 12 | 3 | 28
  >40 years | 86 | 43 | 85 | 48 | 262
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 44 | 87 | 41 | 255
  Male | 22 | 7 | 16 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Disease Index© Questionnaire Score
Description: The Ocular Surface Disease Index© Questionnaire is a 12-item survey assessing the overall severity of dry eye disease per patient. Each question is rated on a 5-point scale ranging from 0=none of the time to 4=all of the time for a total possible score of 0=No disease to 100=Maximum severity of disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Number analyzed (Participants) | 105 | 51 | 103 | 56
Score on a scale
  Baseline | 41.48 (14.797) | 38.27 (12.825) | 40.28 (13.509) | 40.18 (13.443)
  Change from baseline at Day 30 | -15.66 (14.717) | -9.78 (17.986) | -14.59 (15.090) | -13.77 (16.112)

2. Secondary Outcome: Change From Baseline in Tear Break-up Time
Description: Tear Break-up Time (TBUT) was assessed at Baseline and Day 30. TBUT is the time in seconds required for dry spots to appear on the corneal surface after blinking. The shorter the tear break-up time, the worse the dry eye. The worse eye at baseline is used to calculate the change at Day 30. A positive change from baseline indicates improvement.
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Number analyzed (Participants) | 105 | 51 | 103 | 56
Seconds
  Baseline | 4.92 (1.790) | 4.61 (1.739) | 4.94 (1.808) | 5.06 (1.699)
  Change from baseline at Day 30 | 1.36 (2.848) | 1.21 (2.521) | 1.33 (2.497) | 1.06 (2.018)

3. Secondary Outcome: Change From Baseline in Corneal Staining
Description: The cornea is the transparent front part of the eye which covers the iris and pupil. Corneal staining following administration of fluorescein dye in the eye is graded using a 6-point scale (0= no staining, 5 = severe staining) over 5 areas of the clear central part of the eye for a minimum score of 0 and a maximum score of 25. The higher the grade score, the worse the dry eye condition. The worse eye at baseline is used to calculate the change at Day 30. A negative number change from baseline represents a decrease in corneal staining (improvement).
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Number analyzed (Participants) | 105 | 51 | 103 | 56
Score on a scale
  Baseline | 4.9 (3.84) | 5.0 (3.76) | 5.0 (3.92) | 4.7 (3.24)
  Change from baseline at Day 30 | -0.7 (2.90) | 0.1 (3.17) | -1.5 (2.37) | -1.4 (2.89)

4. Secondary Outcome: Change From Baseline in Conjunctival Staining
Description: The conjunctiva is the clear membrane covering the white surface of the eye. Conjunctival staining following ocular administration of lissamine green dye was graded using a 6-point scale (0=no staining, 5=severe staining) over 6 areas of the white part of the eye for a minimum score of 0 and a maximum score of 30. The higher the score, the worse the dry eye condition. The worse eye at baseline is used to calculate the change at Day 30. A negative number change from baseline represents a decrease in the severity of conjunctival staining (improvement).
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on as scale
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Number analyzed (Participants) | 105 | 51 | 103 | 56
Score on as scale
  Baseline | 6.7 (5.69) | 6.3 (4.77) | 6.1 (4.41) | 6.7 (5.37)
  Change from baseline at Day 30 | -0.6 (4.17) | 0.5 (3.77) | -1.2 (3.70) | -0.8 (3.70)

5. Secondary Outcome: Change From Baseline in Schirmer Test Results
Description: The Schirmer Test measures the rate of the secretion of tears produced by the eye over 5 minutes. The results indicate the presence of dry eye (Normal = greater than or equal to 10 millimeters (mm) of tears, Dry Eye = less than 10 mm of tears). The smaller the number, the more severe the dry eye. The worse eye at baseline is used to calculate the change at Day 30. A positive number change from baseline indicates an increase in tears (improvement).
Time Frame: Baseline, Day 30
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Number analyzed (Participants) | 105 | 51 | 103 | 56
millimeters
  Baseline | 10.3 (7.37) | 8.4 (7.26) | 10.4 (6.79) | 10.1 (7.60)
  Change from baseline at Day 30 | 1.8 (6.97) | 2.4 (6.30) | 2.0 (6.27) | 2.6 (6.59)

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | Carboxymethylcellulose Based Eye Drop Formulation B | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops | Carboxymethylcellulose Based Lubricant Eye Drops
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/51 | 0/103 | 1/56
Other Adverse Events (participants affected / at risk) | 0/105 | 0/51 | 0/103 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose Based Eye Drop Formulation A (N=105) | Carboxymethylcellulose Based Eye Drop Formulation B (N=51) | Carboxymethylcellulose Preservative-Free Lubricant Eye Drops (N=103) | Carboxymethylcellulose Based Lubricant Eye Drops (N=56)
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.